CLINICAL TRIAL: NCT03452163
Title: Performance Assessment of the Physiological Monitor Device (PMD-200), a Novel Pain Monitor, in Subjects at Neurointensive Care Unit (NICU).
Brief Title: Performance Assessment of the PMD-200 in Subjects at Neurointensive Care Unit
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to support study performance
Sponsor: Medasense Biometrics Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLI-16-03
Record Dates: First submitted 2018-01-21; First posted 2018-03-02 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2020-03

CONDITIONS: Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anesthesia, General (Experimental): Subjects under anesthesia that are expected to stay for at least 24 hours in the ICU/NICU will be monitored by the PMD-200 device. An EEG monitor device will be connected to the patient and display the Spectral Edge Frequency (SEF) signals and values on the subject monitor.
  Interventions: Device: PMD-200; Device: EEG monitor

INTERVENTIONS:
Device: PMD-200 — the patients will be monitored by PMD-200. The technology consists of measurements of a number of nociception-related physiological parameters that corresponds with the autonomic nervous system's response to noxious stimuli, and using the company's proprietary algorithms, 'translating' these measurements into an index that represents the nociceptive response, the NoL™ (Nociception Level) Index. The NoL index is a relative index from 0 to 100, while 0 is "no pain/nociception" and 100 is "extreme pain/nociception".
Device: EEG monitor — An EEG device will be connected to the patient and display the Spectral Edge Frequency (SEF) signals and values on the subject monitor.

SUMMARY:
Performance Assessment of the PMD-200, a Novel Pain Monitor, in Subjects at Neurointensive Care Unit.

DETAILED DESCRIPTION:
The proposed study is design to further demonstrates the performance of the Nociception Level (NoL) Index in neurological impaired anesthetized patients under general anesthesia, by evaluating its response to controlled changes in the levels of noxious stimuli/analgesia, and to correlate the NoL response to the EEG derived pain score. Validating the performance of the NoL Index may provide a tool to monitor the pain/nociception in this population.

In this study, the PI plan to demonstrate that the NoL Index is a continuous index. It is anticipated that a higher level of nociception will correspond to a higher NoL index. On the other hand, it is anticipated that higher levels of analgesic agent for the same noxious stimulus will lead to a lower NoL index.

The participants will be monitored as in a typical ICU and according to the local guidelines by various types of monitoring devices, such as: vital signs, pulse oximeter, Bispectral Index (BIS), Electroencephalography (EEG) etc.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* The subject is under general anesthesia
* The subject have a blood pressure measurement (either arterial or cuff) during the study
* A signed Informed Consent Form (ICF) has been obtain

Exclusion Criteria:

- The subject is constantly agitate or moving a lot

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Correlation between changes in the nociception levels of the subject (NoL Index value) prior and following a noxious stimuli | Through study completion, about one year
  To demonstrate that the NoL Index is correlates with changes in the nociception levels of the subject prior and following a noxious stimuli.

SECONDARY OUTCOMES:
Correlation between changes in the nociception levels of the subject (NoL Index value) to other nociception predictors (HR, NIBP) | Through study completion, about one year
  The NoL values can be correlate to other nociception predictors (e.g heart rate, blood pressure) following a noxious stimuli.
Correlation between the NoL index and the EEG derived pain score | Through study completion, about one year
  To assess the correlation between the NoL index and the EEG derived pain score during arousal response caused by noxious stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Jean Soustiel, Prof., Principal Investigator — Dept. of Neurosurgery Galilee Medical Center, Nahariya, Israel
Locations (1):
- Galil Medical Center, Nahariya, Israel